CLINICAL TRIAL: NCT00381134
Title: Improving Outcomes in Diabetic Nephropathy
Brief Title: Improving Outcomes in Patients With Kidney Disease Due to Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DK063010-04 (completed)
Record Dates: First submitted 2006-09-26; First posted 2006-09-27 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Diabetes; Kidney Disease; Hypertension
Keywords: double-blind; placebo-controlled; nephropathy; blood pressure; urine albumin to creatinine ratio; placebo
MeSH Terms: conditions — Diabetes Mellitus; Kidney Diseases; Hypertension | interventions — Losartan; Spironolactone

INTERVENTIONS:
Drug: losartan 100 mg orally once daily
Drug: spironolactone 25 mg orally once daily
Drug: placebo once orally once daily

SUMMARY:
Kidney disease affects about one out of three people with diabetes mellitus, a common medical problem. Treatment of kidney disease with medications that lower blood pressure can slow the kidney disease but there is no known cure. This study is designed to test the hypothesis that certain combination-based blood pressure lowering regimens (of FDA approved medications) are better than single agent-based regimens for lowering blood pressure and further slowing or preventing progression of this incurable disease

DETAILED DESCRIPTION:
The long-range objective of this project is to prevent progression of diabetic nephropathy, the leading cause of end-stage renal disease (ESRD). In most patients diabetic nephropathy progresses inexorably to ESRD despite inhibition of the renin-angiotensin- aldosterone system with angiotensin converting enzyme inhibitors (ACEIs) or angiotensin II type 1 receptor blockers (ARBs). The specific aims of this proposal are to: 1) recruit a multiethnic cohort of 78 young adults (ages 20-40) with type 1 (n=36) or type 2 (n=36) diabetes and overt nephropathy (defined as a urine albumin/creatinine ratio > 300 mg albumin/g creatinine) and randomize in a double blind fashion to a control group consisting of ACEI-based therapy alone (ramipril 40 mg once daily) or one of two experimental groups: a) ACEI + ARB (ramipril 40 mg once daily plus losartan 100 mg once daily) or b) ACEI + mineralocorticoid receptor antagonist (MRA) (ramipril 40 mg once daily plus spironolactone 25 mg once daily); 2) conduct a 12-month prospective study to determine if proteinuria is reduced to a greater extent when either the ARB or MRA is added to ACEi-based therapy. This study is powered to detect a 30% greater reduction in 24-hour urine albumin/creatinine ratio in either experimental group versus control (alpha = 0.05, beta=0.10, repeated measures analysis of variance). Secondary endpoints to be examined include: (a) serum potassium and creatinine to assess safety, (b) TGF-beta, as a surrogate marker for ongoing renal injury, (c) plasma renin activity, angiotensin II and aldosterone levels and (d) plasma lipids and lipoprotein composition; and 3) perform repeated ambulatory blood pressure monitoring (ABPM) to examine the renoprotective effect of the 3 different regimens at comparable 24-hour BP of < 125/75 mmHg. The deliverables include: 1) documentation of the safety of maximal dose combination therapy; 2) the feasibility of utilizing 24-hr ABPM to establish BP independent renoprotective effects of specific antihypertensive therapies; and 3) provide preliminary data for future large-scale studies to test efficacy and safety of combining ACEi with MRA therapy on renal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female subjects aged 20-65 of all ethnic backgrounds.
* Type I diabetes mellitus defined as sudden onset of insulin requiring diabetes prior to age 20 and at least 5 years duration
* Type 2 diabetes mellitus defined as onset > 20 years of age and treatment with oral hypoglycemic agent and/or insulin and increased C-peptide level.
* Seated SBP > 130 mmHg documented at one screening visit or treated SBP < 130 mmHg with a documented history of SBP > 130 mmHg on more than one previous occasion
* Proteinuria defined as a 24-hour urine albumin/creatinine ratio > 300 mg/g while on an ACE inhibitor with or without non-ARB, non-aldosterone antagonist treatment
* Ongoing treatment (> 3 months) with an ACE inhibitor or ARB with or without additional antihypertensive therapy (e.g. CCB, a-blocker, b-blocker, clonidine).

Exclusion Criteria:

* BMI > 45 kg/m2
* Baseline serum creatinine > 3.0 mg/dl in females and > 4.0 mg/dl in males or creatinine clearance <20 ml/min estimated by Cockcroft-Gault equation (based on age, fasting serum creatinine concentration and ideal body weight in kilograms).
* Secondary cause of kidney disease other than diabetic nephropathy
* Serum potassium concentration >5.5 mEq/L on ACE inhibitor therapy 7-10 days prior to randomization
* Poorly controlled diabetes, i.e. HgbA1C > 11 mg/dl 7-10 days prior to randomization
* History of allergy to iothalamate or history of renal failure due to contrast nephropathy
* Stroke or myocardial infarction within the preceding 12 months prior to randomization
* Coronary revascularization procedure within past 6 months
* Clinically apparent congestive heart failure defined as clinical signs of heart failure or an ejection fraction of < 40% (and/or depressed LV systolic function by echocardiogram).
* Terminal disease including cancer and AIDS
* Documented increase in serum creatinine > 50% of baseline within 3 months prior to the run-in period
* Renal disease known or in the opinion of the investigator caused by a condition other than diabetes
* Known adverse reaction to study medications including ACE inhibitors, ARB and spironolactone
* History of chronic or intermittent gross hematuria
* Spontaneous 24-hour urine sodium excretion rate exceeding 350 mEq/day
* AST or ALT greater than 2.5 the upper limit of normal for the laboratory
* Pregnancy
* History of autoimmune disease, connective tissue disease or multiple drug allergies
* Anticipated need for renal replacement therapy within 12 months Inclusion criteria for normal subjects
* Adult male and female subjects aged 20-65 of all ethnic backgrounds Exclusion criteria for normal subjects
* Chronic medical conditions, including but not limited to diabetes mellitus, hypertension, chronic kidney disease, and hyperlipidemia.
* Use of medications for antihypertensive
* Inability to follow study protocol for any reason

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2003-07; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Change in 24 hour urine albumin to creatinine ratio after 12 months of treatment

SECONDARY OUTCOMES:
Changes in:
urine transforming growth factor beta
plasma lipids
lipoprotein levels
plasma aldosterone level

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Toto, MD, Principal Investigator — The University of Texas Southwestern Medical Center Dallas
Locations (1):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Natale P, Palmer SC, Navaneethan SD, Craig JC, Strippoli GF. Angiotensin-converting-enzyme inhibitors and angiotensin receptor blockers for preventing the progression of diabetic kidney disease. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD006257. doi: 10.1002/14651858.CD006257.pub2. PMID 38682786
- [Derived] Crompton M, Ferguson JK, Ramnath RD, Onions KL, Ogier AS, Gamez M, Down CJ, Skinner L, Wong KH, Dixon LK, Sutak J, Harper SJ, Pontrelli P, Gesualdo L, Heerspink HL, Toto RD, Welsh GI, Foster RR, Satchell SC, Butler MJ. Mineralocorticoid receptor antagonism in diabetes reduces albuminuria by preserving the glomerular endothelial glycocalyx. JCI Insight. 2023 Mar 8;8(5):e154164. doi: 10.1172/jci.insight.154164. PMID 36749631
- [Derived] Chung EY, Ruospo M, Natale P, Bolignano D, Navaneethan SD, Palmer SC, Strippoli GF. Aldosterone antagonists in addition to renin angiotensin system antagonists for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2020 Oct 27;10(10):CD007004. doi: 10.1002/14651858.CD007004.pub4. PMID 33107592
- [Derived] Srivastava A, Adams-Huet B, Vega GL, Toto RD. Effect of losartan and spironolactone on triglyceride-rich lipoproteins in diabetic nephropathy. J Investig Med. 2016 Aug;64(6):1102-8. doi: 10.1136/jim-2016-000102. Epub 2016 Jul 7. PMID 27388615
- [Derived] Van Buren PN, Adams-Huet B, Nguyen M, Molina C, Toto RD. Potassium handling with dual renin-angiotensin system inhibition in diabetic nephropathy. Clin J Am Soc Nephrol. 2014 Feb;9(2):295-301. doi: 10.2215/CJN.07460713. Epub 2014 Jan 9. PMID 24408116